CLINICAL TRIAL: NCT04459728
Title: KickStart30: A 30-Day Nursing Wellness Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-05-0084
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Substance Use
Keywords: Substance Use, Registered Nurses, Wellness Programs
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness Intervention (Experimental): KickStart30 is an integrated, prescriptive, and trackable wellness intervention combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition.
  Interventions: Behavioral: Wellness Element 1: Exercise; Behavioral: Wellness Element 2: Mindfulness; Behavioral: Wellness Element 3 - Sleep Hygiene; Behavioral: Wellness Element 4 - Social Connectedness; Behavioral: Wellness Element 5 - Nutrition; Behavioral: Wellness Element 6 - Wellness Exercises; Behavioral: Wellness Element 7 - Motivational Messages

INTERVENTIONS:
Behavioral: Wellness Element 1: Exercise — Daily wellness element focusing on Exercise; adherence documented online daily
Behavioral: Wellness Element 2: Mindfulness — Daily wellness element focusing on Mindfulness Meditation; adherence documented online daily
Behavioral: Wellness Element 3 - Sleep Hygiene — Daily wellness element focusing on sleep hygiene; adherence documented online daily
Behavioral: Wellness Element 4 - Social Connectedness — Daily wellness element focusing on social connectedness; adherence documented online daily
Behavioral: Wellness Element 5 - Nutrition — Daily wellness element focusing on nutrition; adherence documented online daily
Behavioral: Wellness Element 6 - Wellness Exercises — Daily wellness workbook exercises focusing on improving mental wellness; adherence documented online daily
Behavioral: Wellness Element 7 - Motivational Messages — Daily motivational emails offering information on one of the 5 wellness elements each day (Exercise, Mindfulness Meditation, Sleep, Social Connectedness, and Nutrition)

SUMMARY:
This study explores the efficacy and feasibility of a self-management wellness intervention that is integrated, prescriptive, and trackable in a population of registered nurses in the state of Texas enrolled in the TExas Peer Assistance Program for Nurses (TPAPN). This 30-day wellness intervention (called "KickStart30") combines five wellness elements: exercise,mindfulness, sleep, social connectedness, and nutrition. Additionally, the program requires that participants implement 5 wellness interventions daily for the 30-day study, document daily online adherence, complete daily HERO (happiness, enthusiasm, resilience, and optimism) exercises to improve mental wellness, and complete online program forms before and after the 30-day intervention. Participants are assessed pre- and post-intervention to determine whether the intervention promotes wellness behavior changes.

DETAILED DESCRIPTION:
TPAPN is a voluntary program funded by the Texas Board of Nursing that provides early identification, support, monitoring, and accountability to Texas nurses who have an identified substance use and/or mental health condition or related incident. The goal of TPAPN is to help the nurse return to safe nursing practice. Currently, TPAPN does not offer a wellness intervention as part of their services. The purpose of this study is to explore the efficacy and feasibility of a self-management wellness intervention that is integrated, prescriptive, and trackable in a population of Texas nurses referred to a peer assistance monitoring program for an identified substance use and/or mental health condition or related incident. It is expected that this 30-day integrated, prescriptive, and trackable wellness intervention (combining five wellness elements including exercise, mindfulness, sleep, social connectedness, and nutrition) will be found to be an efficacious program for those with nurses enrolled in TPAPN.

Nurses are more susceptible to maladaptive coping behaviors, including turning to substance use or abuse, due to workplace stressors (Jarrad et al., 2018). Participating in a nursing monitoring program may increase stress in an already highly stressful profession; monitoring requirements alone can cause feelings of embarrassment and guilt (Mumba, 2018). It is the hope that adding the KickStart30 program, previously studied in a population with mental health issues (Rolin et al., 2019; NCT03993548) to the current offerings of TPAPN will result in the nurse replacing negative coping mechanisms with the positive coping mechanism, increasing long-term recovery and decreasing the likelihood of making an error in the workplace.

To the best of our knowledge, even though there is abundant research supporting each of the KickStart30 elements (exercise, mindfulness, sleep, social connectedness, and nutrition) individually, there is no research exploring the effectiveness of an integrated, prescriptive, and trackable wellness intervention combining these five elements specific to a cohort of nurses. Therefore, this work will be unique in that it will collect both objective and subjective data to assess the feasibility and effectiveness of this type of wellness intervention. It will lend support to the growing body of research on the efficacy of wellness interventions for a variety of different health conditions, as well as a community-based population. Finally, it is hoped that positive results will yield increased access to and utilization of this type of intervention, thereby improving public health.

The recruitment period will be open for 12 months to obtain a maximum of 50 participants. The study population will be nurses, ages 18 and older, interested in improving their overall wellness as part of the TPAPN program. Potential participants will be recruited via TPAPN Case Managers, Peer Support Partners, and Program Director who will provide recruitment flyers to potential participants. The study flyer will be posted to the TPAPN website as well as a informational video for potential participants to view. Interested individuals will be provided a toll-free phone number belonging to study personnel, which will be monitored daily Monday through Friday. Study personnel will reply to interested parties with a verbal screening/orientation call to determine eligibility. If the participant meets study criteria, the participant will be emailed a link to the online consent form, registration form, and program forms. Participants will have the option to download a PDF of their signed consent form for their records at the time of signing/completion. Study personnel will collect the participant's email address, physical mailing address, and assign the participant a unique identification code based on the order in which the participant was screened

Study personnel will mail each participant a KickStart30 Workbook within one day of emailing participants their unique identification codes. Participants will be instructed to document adherence of their daily wellness practices and their daily HERO exercises online via Qualtrics, an online survey software. Participants can document their daily adherence using their computer and/or their smartphone as Qualtrics offers a mobile version of the Participant Tracking Form. A copy of the Participant Tracking Form will also be available in the KickStart30 Workbook so participants that prefer keeping a daily paper log can do so, and they can then transfer their program adherence information to the online Participant Tracking Form at their convenience throughout the program. The workbook will contain the participant's personal identification code; no personal identification will appear in the workbook in order to protect participant confidentiality. Participants will also receive daily motivational emails from MailChimp, which will provide general information about one of the five wellness elements and/or one of the HERO wellness traits, as well as encouragement to track their participation on a daily basis, and encouragement to contact study personnel via email with any questions and/or concerns.

Data capture will occur at two points: once prior to beginning the study and again at the end of the 30-day study. Data will be collected online through program forms; all data will be hosted on Qualtrics, an online survey software. Program Forms assess items including depression, anxiety, wellbeing, mindfulness, sleep quality, social connectedness, emotional eating, pain, disability, physical function, cognition, substance and alcohol use, suicidality, happiness, enthusiasm, resilience, and optimism.

Descriptive statistics will be used to discuss pre- and post-intervention scores.

Differences between pretest and 30-day measures will be assessed with repeated measures ANOVA, with a p value of less than 0.05 indicating statistical significance.

ELIGIBILITY:
Inclusion Criteria:

Licensed nurse in Texas Enrolled in TPAPN services/programs English-speaking Access to a reliable Internet-enabled computer Basic computer skills

Exclusion Criteria:

Acutely suicidal and/or actively psychotic Non-English speaking Participants that are pregnant or plan to get pregnant during the next 30- days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Change in HERO Wellness Scale | 0, and 30 days
  Brief scale that measures 4 wellness traits plus perceived mental wellness

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | 0, and 30 days
  The PHQ-9 is a nine-item depression self-report questionnaire for screening and measurement of severity of major depression. Scores range from 0-27 (lower scores = less depression)
Change in Generalized Anxiety Disorder-7 (GAD-7) | 0, and 30 days
  The GAD-7 is a seven-item self-report questionnaire for screening and measurement of severity of generalized anxiety disorder. Scores range from 0-21 (Lower scores = Less anxiety).
Change in World Health Organization Well-Being Index (WHO-5) | 0, and 30 days
  The WHO-5 Well-Being Index is a five-item self-report questionnaire covering 5 areas: positive mood, vitality, and general interests. Scores range from 0-25 (Higher scores = Higher levels of well-being)
Change in the Short Inventory of Problems Revised (SIP-R), | 0, and 30 days
  a 17-item inventory of adverse consequences associated with drug and alcohol use
Change in Patient Safety Screener (PSS-3) | 0, and 30 days
  a 3-item screening tool for suicidality
Change in the Mindful Attention Awareness Scale (MAAS), | 0, and 30 days
  a measure to assess mindfulness
Change in the Sleep Condition Indicator (SCI), | 0, and 30 days
  a brief scale that assesses for insomnia disorder
Change in the Social Connectedness Scale (SCS), | 0, and 30 days
  a brief scale that assesses social connectedness
Change in the Eating and Appraisal Due to Emotions and Stress (EADES) | 0, and 30 day
  an assessment of utilizing stress and coping skills in relation to food and eating utilizing stress and coping skills in relation to food and eating.
Change in Brief Pain Inventory (BPI) | 0, and 30 days
  a measurement tool for assessing clinical pain.
Change in the Sheehan Disability Scale (SDS), | 0, and 30 days
  a measurement tool for assessing functional impairment in three interrelated domains (work/school, social and family life.)
Change in the Cognitive and Physical Functioning Questionnaire (CPFQ) | 0, and 30 days
  a brief scale that measures cognitive and executive dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Saundra M Jain, PsyD, LPC, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jarrad R, Hammad S, Shawashi T, Mahmoud N. Compassion fatigue and substance use among nurses. Ann Gen Psychiatry. 2018 Mar 13;17:13. doi: 10.1186/s12991-018-0183-5. eCollection 2018. PMID 29563960
- [Result] Mumba MN. Employment implications of nurses going through peer assistance programs for substance use disorders. Arch Psychiatr Nurs. 2018 Aug;32(4):561-567. doi: 10.1016/j.apnu.2018.03.001. Epub 2018 Mar 7. PMID 30029748
- [Result] Rolin D, Fox I, Jain R, Cole SP, Tran C, Jain S. Wellness Interventions in Psychiatrically Ill Patients: Impact of WILD 5 Wellness, a Five-Domain Mental Health Wellness Intervention on Depression, Anxiety, and Wellness. J Am Psychiatr Nurses Assoc. 2020 Sep/Oct;26(5):493-502. doi: 10.1177/1078390319886883. Epub 2019 Nov 18. PMID 31738111